CLINICAL TRIAL: NCT04697823
Title: Effect of Hyaluronan-enriched Medium on the Cumulative Ongoing Pregnancy Rate: a Prospective Randomized Trial
Brief Title: Effect of Hyaluronan-enriched Medium on the Cumulative Ongoing Pregnancy Rate.
Acronym: TETHER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Sophie Debrock, clinical embryologist, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S64387
Record Dates: First submitted 2020-12-16; First posted 2021-01-06 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hyaluronan-EnRiched Medium; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Patients receiving an embryo transfer in hyaluronan-enriched transfer medium
  Interventions: Other: use of hyaluronan-enriched transfer medium
- control group (No Intervention): Patients receiving an embryo transfer in conventional culture medium

INTERVENTIONS:
Other: use of hyaluronan-enriched transfer medium — In the study group, an embryo transfer will be performed in hyaluronan-enriched transfer medium
  Arms: study group

SUMMARY:
Assessing whether the use of hyaluronan-enriched transfer medium can increase the cumulative ongoing pregnancy rate

ELIGIBILITY:
Inclusion Criteria:

* Patients with own oocytes/embryos;
* Patients with female age at 1st OR in the study <40 year;
* Patients planned for a 2nd oocyte retrieval, with no clinical ongoing pregnancy after the previous oocyte retrieval
* Patients planned for a 3rd oocyte retrieval with no clinical ongoing pregnancy after previous oocyte retrievals
* Patients with female age at 1st OR in the study <40 year;
* Patients with BMI ≤32;
* Patients with written informed consent;

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
number of transfers needed to reach ongoing pregnancy | ongoing defined as a pregancy with a viable fetus with FHB at 12 weeks of pregnancy
  The primary outcome parameter is the number of transfers needed to reach ongoing pregnancy (ongoing defined as a pregancy with a viable fetus with FHB at 12 weeks of pregnancy), as a time-to-event outcome variable. Patients that do not reach pregnancy, are censored at their last transfer.

SECONDARY OUTCOMES:
number of transfers needed to reach clinical pregnancy, life birth, miscarriage, multiple pregnancy | until Live birth: 9 months after ET
  clinical pregnancy is defined as a pregnancy with at least one intrauterine (IU) or extrauterine (EU) fetal sac at 6-7 weeks of pregnancy)

CONTACTS AND LOCATIONS:
Locations (1):
- Leuven University Fertility Center, Leuven, Belgium